CLINICAL TRIAL: NCT04148547
Title: Transcranial Direct Current Stimulation (tDCS) in the Primary Motor Cortex and Its Effects on Sensitivity, Pressure Pain Threshold, and Electromyographic Activity in Healthy Individuals: A Quasi-experimental Single-blind Sham-controlled Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) in the Primary Motor Cortex in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: uammadrid4
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Basic Physiology; Brain Stimulation
Keywords: Transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial direct current stimulation (Experimental)
  Interventions: Device: Sooma transcranial direct current stimulation device
- Sham transcranial direct current stimulation (Placebo Comparator)
  Interventions: Device: Placebo Sooma transcranial direct current stimulation device

INTERVENTIONS:
Device: Sooma transcranial direct current stimulation device — This group received brain training through transcranial direct current for 20 minutes.
  Arms: transcranial direct current stimulation
Device: Placebo Sooma transcranial direct current stimulation device — This group received sham brain training through transcranial direct current for 20 minutes. The current is active for 15 seconds and then switches off until the intervention is finished.
  Arms: Sham transcranial direct current stimulation

SUMMARY:
The main aim of this study is to assess the short-term effects of active-tDCS (a-tDCS) on the M1 regarding sensorimotor variables such as discriminative sensation, pressure pain threshold and electromyographic activity compared with a sham-tDCS (s-tDCS) in healthy individuals. The main objective was to determine whether there were clinically relevant changes generated by tDCS and if they were superior to a sham intervention.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic participants
* men and women aged 18 to 65 years

Exclusion Criteria:

* insomnia
* nausea
* headache
* pregnancy
* use of painkillers in the last 24 hours
* presence of metal inside the head
* pacemaker
* wound on the area of electrodes' application
* drug consumption; (j) recent application of tDCS
* psychiatric disease impeding understanding of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold through an algometer | Change in pressure pain threshold immediately at the end of the intervention
  Pressure pain threshold has been defined as the minimal amount of pressure at which a sense of pressure first changes to pain or discomfort
Tactile acuity threshold | Change in tactile acuity threshold immediately at the end of the intervention
  Tactile acuity threshold is an important variable to know the somatosensory state and Von Frey monofilaments and Aesthesiometer were used
Muscle recruitment through electromyographic activity | Change in electromyographic activity immediately at the end of the intervention
  The activity of surface electromyography (sEMG) during an isometric maximal voluntary contraction was measured in the biceps brachii and rectus femoris.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No